CLINICAL TRIAL: NCT06641726
Title: Developing an Internationally-diverse, Linked Genomic and Longitudinal Phenotypic Research Dataset to Accelerate Precision Psychiatry for Patients With Serious Mental Illness
Brief Title: Creating a Global Research Database That Connects Genetic Information and Long-term Health Data to Improve Personalized Treatment for People With Serious Mental Illness
Acronym: GlobalMinds
Status: Recruiting | Type: Observational
Sponsor: Akrivia Health (Industry)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: GM001; 328854 (Other: IRAS)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder (BD); Schizophrenia Disorders; Major Depressive Diorder; Dementia
Keywords: cross-sectional; observational; bioresource; biomarkers; whole genome sequencing; linked bioresource; dementia; neuropsychiatric
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — Extracted DNA samples, plasma, serum and derived PBMCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: 40,000 participants with linked EHR and baseline assessments will provide a DNA sample only, via saliva or blood. This cohort will comprise even distribution across neuropsychiatric disorders including Schizophrenia, Major depressive disorder (MDD), and Bipolar diagnostic groups (approximately 13,300 patients in each group).
  Interventions: Other: Not applicable- observational study
- Cohort 2: 9,000 participants with linked EHR and baseline assessments patients will provide DNA, RNA, peripheral blood mononuclear cells (PBMCs), plasma and serum via blood. This cohort will also comprise even distribution across neuropsychiatric disorders including Schizophrenia, Major depressive disorder (MDD), and Bipolar diagnostic groups (approximately 3000 patients in each group).
  Interventions: Other: Not applicable- observational study
- Cohort 3: 1000 participants with Dementia who have linked EHR and assessments will provide DNA, RNA, peripheral blood mononuclear cells (PBMCs), plasma and serum via blood.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — This is non-interventional, cross-sectional observational study and thus there is no intervention.

SUMMARY:
This observational study aims to provide new insights into the nature and classification of severe mental illness and dementias that in time should help improve diagnostic practise, and enable the development of new and improved treatments. The investigators will achieve aims by gathering information and biological samples from over 50,000 research participants and then linking this information with participants' electronic health records, genetic and other potential markers of mental illnesses (called biomarkers, derived from biological samples). The investigators will use this resource to analyse how potential risk factors - genetic, other biological and non-biological (related to the participants' life circumstances) - influence participants' experiences, symptoms, and outcomes (both mental and physical health). The investigators will also use advanced analysis to assess whether there may be better ways of grouping together and understanding the experiences of those with severe mental illnesses and dementias. Given the value and importance of this resource for advancing mental health research, the investigators will also make the data available to other researchers to pursue these broad research aims.

DETAILED DESCRIPTION:
GlobalMinds is a research study with the goal of creating a precision psychiatry bioresource combining biological and clinical data on 50,000 participants with severe mental illness and dementia. The investigators will use this resource to investigate how genomics, other biological measures and non-biological risk factors are associated with these conditions and their outcomes. In addition, the investigators will deploy advanced analytic approaches to explore whether the combined dataset can help us derive more precise classification and diagnostic approaches and better prediction of outcomes. The investigators will also work with other researchers and enable access to the dataset to address these questions. In doing so, the investigators seek to enable the development of novel treatment options and improved, biologically informed classification for the most challenging conditions in psychiatry and dementia.

The GlobalMinds programme is a precision neuroscience initiative (PNI). Its purpose is to improve the quality and availability of genomic and health care data for research into severe neuropsychiatric and degenerative ilnesses . The study will involve the whole genome sequencing from 50,000 patients suffering from neuropsychiatric and neurodegenerative disorders and linking this data to their individual electronic health records (EHRs) available within the Akrivia Health platform.

No investigational product will be used, but the trial will deploy methods of clinical phenotyping, genomic sequencing, biobanking, diverse recruitment strategies in order to allow researchers to identify translatable biomarkers and disease-modifying targets for drug development downstream.

This research study will develop a recruitment infrastructure that embraces the advantages conferred by the NHS research ecosystem, but crucially adds to existing NIHR and NHS strategies in order to meet our ambitious recruitment target. In GlobalMinds a national multi-media participant engagement campaign, delivered in partnership with the NHS, will direct patients with capacity to a centralised digital portal - the GlobalMinds Hub - to automate a large proportion of study activity. This process will be managed by a dedicated study team run by Akrivia Health. The GlobalMinds study team will monitor recruitment rates and sample diversity, provide quality assurance on participant-generated data, coordinate the network of expert project partners responsible for the national engagement campaign, PPI, and digital infrastructure, and crucially undertake local community outreach, targeted recruitment and in-person sample collection to minimise the risk of digital exclusion. For 40,000 participants who will provide DNA for whole genome sequencing, patients will be screened and recruited into the study remotely and issued a remote DNA capture pack that patients can use and return in their own time. Where participants express an interest in doing so, on-site and mobile phlebotomy services will be used to obtain bloods samples for participants electing to participate in the biomarker cohort.

The investigators will use the Global Minds data resource to address broad research objectives, but also work with, and provide secure access to the data resource, for the wider research community, both academic and non-academic researchers in the UK and abroad. Levels of access will be determined by Akrivia's Data Access Committee upon request from a research team.

ELIGIBILITY:
Inclusion Criteria:

- All participants must have an electronic health record in a primary or secondary care service.

Mental Health cohort(s) • Have received a diagnosis and/or treatment/referral for mental illness for MDD, BD, Schizophrenia.

• Having an available electronic health record

• Current age 18+ (no upper age limit)

• Can speak English Dementia cohort

• Participants aged 18+ (no upper age limit)

• Currently alive and are, or have been, old age psychiatry patients

•

Received relevant diagnosis or referral:

EITHER

• Clinical diagnosis of dementia, mild cognitive impairment (MCI) or subjective cognitive impairment (SCI) OR

• Memory clinic referral

• Must be willing and able to complete a validated cognitive assessment (MoCA or SLUMS).

All dementia patients will undergo the extended biomarker analysis.

Exclusion Criteria:

- Mental Health cohort(s)

• Patients without capacity to provide consent. Dementia cohort

• Inability to understand spoken and/or written spoken English

• Individuals with intellectual disability.

• Patients with dementia in Creutzfeldt-Jakob disease (CJD), Huntington's, HIV dementia, alcohol-related dementia, intellectual disability, traumatic brain injury at any time.

• Patients diagnosed with depression (only an exclusion criterion for MCI/SCI patients), psychosis, bipolar disorder prior in the pre-index period - to be checked at screening.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 and over with neuropsychiatric (MDD, BD or Schizophrenia) or Neurodegenerative disorder (dementia).
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of participants with schizophrenia, bipolar disorder or schizoaffective disorder | 1 month from sample collection and baseline assessment.
  The primary outcome measure of this study is the diagnosis of participants with bipolar disorder, schizophrenia or schizoaffective disorder in accordance with ICD-10 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Prof. James Walters, Principal Investigator — Cardiff University
Locations (1):
- GlobalMinds central study team, Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be shared with researchers at the discretion of the data access committee, but no individual identifiable patient data will be shared.